CLINICAL TRIAL: NCT00848809
Title: Pharmacokinetics of Vancomycin in Various Modalities of Renal Replacement Therapy in the Intensive Care Unit
Brief Title: Pharmacokinetics of Vancomycin in the ICU in Renal Replacement Therapy
Status: Withdrawn | Type: Observational
Why Stopped: PI had difficult enrollment.
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Bradley Beck, Pharm.D., Avera McKennan Hospital and University Health Center
Other Study IDs: 2008.073
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Vancomycin therapy; Slow-low efficiency daily dialysis; Intermittent Hemodialysis; Kidney; Vancomycin; Hemofiltration
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection; Vancomycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Slow-low efficiency daily dialysis group
  Interventions: Procedure: Blood sample
- 2: Intermittent Hemodialysis group
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — 9 blood samples will be sent to the laboratory for the subjects in the SLED cohort
  Other Names: Vancomycin level
  Groups: 1
Procedure: Blood sample — 10 blood samples will be collected and sent to the laboratory for the subjects in the intermittent hemodialysis cohort.
  Other Names: Vancomycin level
  Groups: 2

SUMMARY:
This study is an observational analysis that monitors the effect of different dialysis methods on vancomycin levels when patients are critically ill. No changes are made to therapy based on levels, but levels are checked more frequently than normal. The primary dialysis methods being studied are SLED (slow-low efficiency daily) dialysis and intermittent hemodialysis. Vancomycin is the only medication being evaluated in this study. This study will provide detailed information on how to dose vancomycin in patients that are on dialysis in the intensive care unit.

DETAILED DESCRIPTION:
The proposed study will evaluate the pharmacokinetics of vancomycin in patients that are on being treated with various types of renal replacement therapy. The renal replacement therapies studied in this trial will be slow-low efficiency daily (SLED) dialysis and intermittent hemodialysis. This data will be collected and plotted for vancomycin for each dialysis mechanism utilized and plotted on drug concentration versus time graphs to determine drug clearance in each type of renal replacement therapy. Subjects will have blood samples drawn and sent to the laboratory according to the dialysis method studied (9 for SLED dialysis and 10 samples for intermittent hemodialysis). Serial levels will be drawn prior to the drug being administered and after the drug is infused to assess the clearance and distribution of vancomycin. Study drug levels will be drawn from blood that is already available in the laboratory when timing of such samples is appropriate, in order to limit the amount of blood that is drawn from each study subject. A total of 30 milliliters of blood will be collected from each subject for any one study arm they fit into. Blood will be collected no more than two times per week and only more than once in a particular patient if their dialysis regimen changes. A single particular subject will only be able to supply blood samples once for each dialysis regimen being studied. This study would allow for the data collection of vancomycin levels at several time points during renal replacement therapy to assess the pharmacokinetic parameters associated with vancomycin dosing in each specialized patient-dialysis combination.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* One of the following types of dialysis modalities implemented:

Slow-low efficiency daily dialysis Intermittent hemodialysis

* Use of study medication (vancomycin)

Exclusion Criteria:

* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be admitted to the intensive care unit at Avera McKennan Hospital in Sioux Falls, SD.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the effect of different types of renal replacement therapies on the elimination and volume of distribution of vancomycin. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Beck, Pharm.D., Principal Investigator — Avera McKennan Hospital and University Health Center
Locations (1):
- Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Kielstein JT, Czock D, Schopke T, Hafer C, Bode-Boger SM, Kuse E, Keller F, Fliser D. Pharmacokinetics and total elimination of meropenem and vancomycin in intensive care unit patients undergoing extended daily dialysis. Crit Care Med. 2006 Jan;34(1):51-6. doi: 10.1097/01.ccm.0000190243.88133.3f. PMID 16374156
- [Background] Trotman RL, Williamson JC, Shoemaker DM, Salzer WL. Antibiotic dosing in critically ill adult patients receiving continuous renal replacement therapy. Clin Infect Dis. 2005 Oct 15;41(8):1159-66. doi: 10.1086/444500. Epub 2005 Sep 12. PMID 16163635
- [Background] Pai AB, Pai MP. Vancomycin dosing in high flux hemodialysis: a limited-sampling algorithm. Am J Health Syst Pharm. 2004 Sep 1;61(17):1812-6. doi: 10.1093/ajhp/61.17.1812. PMID 15462252